CLINICAL TRIAL: NCT06684106
Title: Ursodeoxycholic Acid Attenuates Statin-Induced Impaired Glucose Tolerance: A Randomized Controlled Clinical Trial
Brief Title: Ursodeoxycholic Acid Attenuates Statin-Induced Impaired Glucose Tolerance
Acronym: URSTAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XJTU1AF2023LSK-149-01; CSCF2022B04 (Other Grant/Funding Number: 2022 Chinese Society of Cardiology's Foundation)
Record Dates: First submitted 2024-11-04; First posted 2024-11-12 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hyperlipidemia; Ursodeoxycholic Acid; Statin Therapy; Glucose Intolerance
MeSH Terms: conditions — Hyperlipidemias; Glucose Intolerance | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ursodeoxycholic acid group (Experimental): Ursodeoxycholic acid (UDCA) 500 mg: This group of participants receive UDCA 500mg per day.
  Interventions: Drug: Ursodeoxycholic acid (UDCA) 500 mg
- placebo group (Placebo Comparator): This group of participants receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ursodeoxycholic acid (UDCA) 500 mg — UDCA together with statin in eligible participants
  Other Names: Ursodeoxycholic Acid; UDCA
  Arms: Ursodeoxycholic acid group
Drug: Placebo — placebo together with statin in ASCVD patients
  Arms: placebo group

SUMMARY:
The purpose of this clinical trial is to understand whether the drug Ursodeoxycholic acid (UDCA) can prevent glucose intolerance in participants with hyperlipidemia who are taking statins. It will also assess the safety of UDCA. The primary questions it aims to answer are:

* Will UDCA reduce the incidence of glucose intolerance in participants taking oral statins?
* Will the use of UDCA decrease other adverse events in patients taking oral statins?

Participants will:

* Take Atorvastatin combined with UDCA or a placebo daily for 6 months
* Have follow-up visits on day 40, day 110, and day 180 Have their examination indicators recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old.
* LDL-C≥3.4mmol/l (130 mg/dL).
* Glycosylated hemoglobin ≤ 6.0% (42 mmol/mol).
* Voluntarily sign informed consent.

Exclusion Criteria:

* Previous diagnosis of diabetes or prediabetes.
* Past or current use of hypoglycemic drugs.
* Oral administration of statin lipid-lowering drugs within three months before enrollment.
* Combined oral drug quantity ≥3.
* History of ASCVD (previous myocardial infarction, ACS, stroke or TIA within 1 year, symptomatic peripheral vascular disease).
* Active liver disease (defined as elevation of alanine aminotransferase (ALT), aspartate aminotransferase (AST) >2 × upper limit of normal (ULN) from any existing known liver infectious, neoplastic, or metabolic pathologic cause or unknown cause at the time of screening), Severe hepatic insufficiency and biliary obstruction.
* Difficult to control hypertension: defined as systolic blood pressure ≥180mmHg or diastolic blood pressure ≥110mmHg despite antihypertensive therapy prior to randomization.
* Estimated glomerular filtration rate (eGFR) ≤ 30 mL/min/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) method
* New York Heart Association (NYHA) Class IV heart failure or a known left ventricular ejection fraction < 25%
* A clinically significant and drug- or ablation-resistant arrhythmia within 3 months prior to randomization
* An acute or severe systemic infection, or any of the following diseases: hematological disorders, autoimmune disorders, malignant tumors, psychiatric patients, or other serious or unstable conditions that could impact study health status
* Scheduled for surgery within 6 months
* Pregnant, breastfeeding, or trying to become pregnant during the study or within 6 months of study completion
* Subjects with alcohol or other drug addiction
* Secondary hypercholesterolemia, such as hypothyroidism or nephrotic syndrome
* A history of allergic reaction to any study drug or its excipients or similar chemical classes of drugs
* A family history of homozygous familial hypercholesterolemia
* Participants currently enrolled in another clinical trial, or who cannot adhere to 6-month follow-up
* Any condition that the investigator considers unsuitable for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-11-11 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 6 months after randomization
  Changes of glycosylated hemoglobin after taking ursodeoxycholic acid for half a year

SECONDARY OUTCOMES:
Concentration of fasting blood glucose | 6 months after randomization
  The concentration of fasting blood glucose was measured and serum was extracted for laboratory testing.
Concentration of fasting islets | 6 months after randomization
  The concentration of fasting islets was measured and serum was extracted for laboratory testing. we use the level of physiological parameter to describe the concentration of fasting islets.
Concentration of blood lipid | 6 months after randomization
  The concentration of blood lipid was measured and serum was extracted for laboratory testing.we use the level of physiological parameter to describe the concentration of blood lipid, including "the level of triglycerides","the level of low-density lipoprotein", "the level of high-density lipoprotein", "the level of total cholesterol" ,"the level of Lipoprotein(a)".
Body composition analysis Fat mass | 6 months after randomization
  The Body composition analysis was measured by the Inbody. we wue the physiological parameter to describe the body composition. e.g."Fat mass"
Body composition analysis Muscle mass | 6 months after randomization
  The Body composition analysis was measured by the Inbody. we wue the physiological parameter to describe the body composition. e.g. "Muscle mass".

CONTACTS AND LOCATIONS:
Overall Officials: Zuyi Yuan, Professor, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (2):
- China (2):
  - Department of Cardiology, First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an

IPD SHARING:
Plan to Share IPD: Undecided